CLINICAL TRIAL: NCT01556555
Title: Prospective Evaluation of the Clinical Utility of Peroral Cholangiopancreatoscopy With the Spyglass System in Patients With Sclerosing Cholangitis
Brief Title: Clinical Utility of the Spyglass System in Primary Sclerosing Cholangitis (PSC)
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Annika Bergquist, Head of department of gastroenterology and hepatology, associate professor, Karolinska University Hospital
Other Study IDs: 552/03
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Sclerosing Cholangitis
Keywords: Sclerosing cholangitis; Spyglass; Endoscopic retrograde cholangiopancreaticography
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary sclerosing cholangitis: Patients with a definite diagnosis of sclerosing cholangitis and a clinical indication for ERCP.

SUMMARY:
This study aim to prospectively evaluate the clinical utility of Spyglass in sclerosing cholangitis patients undergoing endoscopic retrograde cholangiopancreaticography (ERCP). Fifty patients with a definite diagnosis of sclerosing cholangitis and a clinical indication for ERCP from September 2008 and onwards will be investigated with peroral cholangioscopy using Spyglass direct visualization system. Clinical data on all patients will be collected at time of the ERCP including information on the Primary sclerosing cholangitis (PSC) and inflammatory bowel disease (IBD), serum liver function tests and indication for ERCP.

A structured data collection form including information on Majoie Score, macroscopic features of the bile ducts at cholangioscopy, quality of the investigation, technical difficulties, and an overall judgment of whether any abnormalities observed were benign or malignant was completed by the endoscopist in conjunction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* sclerosing cholangitis with indication for ERCP
* Over 18 year
* informed consent

Exclusion Criteria:

* Not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SC, sclerosing cholangitis, who is undergoing ERCP, (Endoscopic Retrograde Cholangio and Pancreaticography)
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annika Bergquist, Assoc prof, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Arnelo U, von Seth E, Bergquist A. Prospective evaluation of the clinical utility of single-operator peroral cholangioscopy in patients with primary sclerosing cholangitis. Endoscopy. 2015 Aug;47(8):696-702. doi: 10.1055/s-0034-1391845. Epub 2015 Mar 31. PMID 25826274